CLINICAL TRIAL: NCT03441464
Title: Feasibility of the LUM Imaging System for Detection of Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim analysis indicated a change in study design to collect in vivo data
Sponsor: Lumicell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL0005
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer; Neoplasm, Residual
Keywords: Fluorescence; Prostate; Cancer detection
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- 1st Tier Dose Level (Experimental): 3 patients administered single dose of LUM015 at 0.5 mg/kg. Imaging with the LUM imaging device will be performed ex vivo on resected tissue.
  Interventions: Combination Product: LUM Imaging System
- 2nd Tier Dose Leel (Experimental): 3 patients administered single dose of LUM015 at 1.0 mg/kg. Imaging with the LUM imaging device will be performed ex vivo on resected tissue.
  Interventions: Combination Product: LUM Imaging System
- 3rd Tier Dose Level (Experimental): After evaluation of the fluorescence signal observed with the LUM imaging device in the three other cohorts,the subsequent 3 patients will receive a dose of 0.5-1.5 mg/kg.
  Interventions: Combination Product: LUM Imaging System
- Auto-fluorescence (No Intervention): No LUM015 injection will be given to three (3) patients to measure baseline tissue fluorescence. The tissue will still be imaged ex-vivo using the LUM Imaging Device

INTERVENTIONS:
Combination Product: LUM Imaging System — Patients will be injected with one of 3 study doses of LUM015, or have no LUM015 intervention, and resected tissue will be imaged ex vivo with the LUM imaging device.
  Arms: 1st Tier Dose Level; 2nd Tier Dose Leel; 3rd Tier Dose Level

SUMMARY:
The primary objective of this feasibility study is to determine if administration of LUM015 will result in positive fluorescence of tumor tissue from ex vivo specimen imaging with the LUM Imaging device from patients undergoing radical prostatectomy for prostate cancer. Both normal tissue and tumor tissue will be imaged and analyzed. The LUM Imaging System is a portable combination product consisting of an imaging device and an imaging agent (LUM015).

Patients with an established diagnosis of prostate cancer and who are eligible for radical prostatectomy will be screened. Eligible patients will be enrolled and on the day of their planned surgery, LUM015 will be administered 2-6 hours prior to surgery. Patients will undergo radical prostatectomy 2-6 hours after LUM015 administration. All surgical specimens will be imaged with the LUM imaging device and have routine diagnostic assessment. Patients will be monitored for adverse events from time of injection through the first standard of care post-surgical follow-up visit.

DETAILED DESCRIPTION:
The primary objective of this feasibility study is to determine if administration of LUM015 will result in positive fluorescence of tumor tissue from ex vivo specimen imaging with the LUM Imaging device from patients undergoing radical prostatectomy for prostate cancer. Both normal tissue and tumor tissue will be imaged and analyzed. The LUM Imaging System is a portable combination product consisting of an imaging device and an imaging agent (LUM015).

Patients with an established diagnosis of adenocarcinoma of the prostate and who are eligible for radical prostatectomy will be screened. Patients will be seen by their surgeon in an office visit and undergo routine preoperative testing within 8 weeks of their planned procedure. After obtaining informed consent and confirming eligibility, patients will be enrolled and on the day of their planned surgery, LUM015 will be administered by bolus intravenous injection 2-6 hours prior to surgery. This injection is the only procedure that will be performed on patients outside of their routine care (standard of care).

LUM015 will be administered in a single dose between 0.5 -1.5 mg/kg in up to 9 patients. An additional 3 patients will not be injected with LUM015, but their specimens will undergo LUM imaging.

Patients will undergo radical prostatectomy 2-6 hours after LUM015 administration. All surgical specimens will be sent to the pathology suite for imaging with the LUM imaging device and routine diagnostic assessment. Imaging will be performed on the resected specimens. Alternatively, specimens can also be imaged in the operating room. Imaged areas showing high fluorescence will be marked with ink to guide pathology evaluation and determine whether the area contains tumor. Samples of imaged areas showing low fluorescence signal will also be evaluated by pathology to determine whether the area only contains normal tissue. Additional resection will not be performed if a positive surgical margin is detected by imaging.

Patients are expected to be admitted to the hospital for the surgical procedure and will remain in the hospital post-surgery per standard of care treatment. Laboratory studies will be performed to assess for any imaging agent related adverse events prior to hospital discharge and at the standard of care post-surgical follow-up visit. Patients will be followed through their first standard of care post-surgical visit. Additionally, patients will be monitored for adverse events from time of injection through the first standard of care post-surgical visit. Patients with adverse events that are possibly related to LUM015 will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically localized or locally advanced prostate cancer and scheduled for radical prostatectomy
* Age 40 years or older
* Able and willing to follow study procedures and instructions
* Received and signed informed consent form
* Otherwise healthy except for diagnosis of cancer
* Normal organ and marrow function as defined below:

  * Hemoglobin 13.9 - 16.3 g/dL
  * Leukocytes 4500 - 11,000 uL
  * Platelets 150,000 - 450,000 uL
  * Total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) within normal institutional limits
  * Creatinine within normal institutional limits or creatinine clearance within normal institutional limits
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Known current substance addiction
* Have taken an investigational drug within 30 days of enrollment
* Received methylene blue prior to tissue excision
* QT Interval > 480ms
* Have not recovered from an adverse event due to pharmaceutical or diagnostic agent
* Uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 100 mm Hg; subjects with known HTN should be under these values while under pharmaceutical therapy
* History of allergic reaction attributed to drugs containing polyethylene glycol (PEG).
* History of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Sexually active subjects unwilling/unable to use medically acceptable forms of contraception during study participation
* HIV-positive subjects on combination antiretroviral therapy
* Investigator feels subject's participation is not in the best interest of the subject
* Previously treated with local or systemic therapies to treat prostate cancer

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with established diagnosis of prostate cancer
Enrollment: 9 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Determine initial efficacy of LUM015 in labeling prostate cancer by molecular imaging by comparing imaging results with pathology | Day 1
  Correlate the fluorescence levels in tumor tissue from ex-vivo specimen imaging to the dose of LUM015 injected.

SECONDARY OUTCOMES:
Number of patients with reported adverse events | Up to 14 days post surgery
  Reported adverse events will be assessed and aggregated according to event type, relation to device or drug, and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Tewari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No